CLINICAL TRIAL: NCT03553524
Title: Time of Day Dependant Effects of High Intensity Interval Training on Blood Glucose Levels in Participants With Type 2 Diabetes
Brief Title: Circadian High Intensity Interval Training Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to personnel and organizational issues.
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Harriet Wallberg, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CircHIIT Study
Record Dates: First submitted 2018-04-13; First posted 2018-06-12 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes; Insulin Independent
Keywords: Type 2 Diabetes; Insulin independent; HIIT; CGM-based blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning first (Experimental): Both arms of the study will perform the baseline measurements during visit 1. Arm 1 of the study will perform HIIT at 08:30 during visit 2, and after a 1-week washout period will perform HIIT at 19:30 during visit 3.
  HIIT bout will consist of 3 minutes of warm-up followed by 6 1-minute intervals of full exertion cycling on a cycle ergometer, interspersed by a 1-minute recovery periods and ending with a 3-minute cooldown.
  Interventions: Other: morning HIIT --> afternoon HIIT
- Afternoon first (Experimental): Both arms of the study will perform the baseline measurements during visit 1. Arm 2 of the study will perform HIIT at 19:30 during visit 2, and after a 1-week washout period will perform HIIT at 08:30 during visit 3.
  HIIT bout will consist of 3 minutes of warm-up followed by 6 1-minute intervals of full exertion cycling on a cycle ergometer, interspersed by a 1-minute recovery periods and ending with a 3-minute cooldown.
  Interventions: Other: afternoon HIIT --> morning HIIT

INTERVENTIONS:
Other: morning HIIT --> afternoon HIIT — Arm 1 will start with morning HIIT at visit 2 and afternoon HIIT at visit 3
  Arms: Morning first
Other: afternoon HIIT --> morning HIIT — Arm 2 will start with afternoon HIIT at visit 2 and morning HIIT at visit 3
  Arms: Afternoon first

SUMMARY:
High intensity interval training (HIIT) is a promising intervention for treatment and prevention of type 2 diabetes. In spite of the interplay between circadian rhythms and exercise, the time of day in which the most robust adaption to HIIT can be achieved is unknown. The main goal of the study is to compare the efficacy of morning and afternoon HIIT in lowering blood glucose values in participants with type 2 diabetes.

DETAILED DESCRIPTION:
High intensity interval training (HIIT) is a promising intervention for treatment and prevention of type 2 diabetes. In spite of the interplay between circadian rhythms and exercise, the time of day in which the most robust adaption to HIIT can be achieved is unknown. The main goal of the study is to compare the efficacy of morning and afternoon HIIT in lowering blood glucose values in participants with type 2 diabetes. Additionally, we aim to to elucidate the underlying hormonal changes and fuel utilization preference responsible for the differing blood glucose response.

A randomized cross-over trial with 40 participants with type 2 diabetes will be performed. The participants will be examined on three occasions on an in-patient basis (36-hour hospital visits). On visit 1 baseline (no exercise) measurements will be established. On visit 2 the participants will perform a single bout of HIIT either in the morning (08:30) or afternoon (19:30). After a 1-week washout period, the participants will return for visit 3 and an opposing exercise time. Primarily, the efficacy of the morning and afternoon HIIT will be judged by the continuous glucose monitor (CGM) -based glycaemia measurements. Additionally, during the visits the investigators will collect repeated blood samples to assess the effect of exercise timing on the diurnal hormonal rhythms. Fuel utilization preference will be measured by respiratory exchange ratio (RER)during exercise.

The hypothesis is that afternoon HIIT will be more efficacious in controlling blood glucose values, based on the preliminary data gathered from the 'free living' pilot study. The current study will aim to compare the morning and afternoon exercise in controlled conditions, eliminating the effects of dietary intake, medication and sleep cycle disruption. Additionally, the specific factors responsible for the differing glycaemic response to morning and afternoon exercise will be elucidated.

Preliminary data from the pilot study

A randomised cross-over pilot study with 11 participants with type 2 diabetes in 'free living' conditions has been performed. Glycaemia measurements were collected by continuous glucose monitors (CGMs) for 2 weeks pre-training and for the duration of the study. The participants were assigned to either morning (08:00) or afternoon (16:00) training regime consisting of 6 HIIT occasions over 2 weeks. Following a 2-week 'wash-out' period, the participants performed the opposing exercise training regime. The preliminary results show that HIIT is more efficacious in improving glycaemia when performed in the afternoon, rather than in the morning.

This pilot was a field-based study in 'free-living' individuals, thus the specific factors responsible for the differing blood glucose levels between morning and afternoon exercise trials remain to be elucidated. Now is the aim to perform a study in controlled condition, limiting the effects food intake, medication and sleep-wake cycle disruption and measuring the effects of a single HIIT bout on glycaemia. The hypothesis is that HIIT bout at different times of day diversely affects diurnal hormonal rhythms, accounting for the differing glycaemic responses.

ELIGIBILITY:
Inclusion criteria

* Age: 45 - 68 years
* Body Mass Index (BMI): 23 - 33 kg/m2
* Participant diagnosed with Type 2 Diabetes (insulin independent)
* Ability to provide informed consent
* Ability to complete the exercise regiment

Exclusion criteria:

* Medications: Insulin
* Current nicotine user (cigarettes, snus, nicotine gum)
* Past nicotine use less than 6 months before inclusion in the study
* Pre-existing cardiovascular condition: Angina pectoris, Cardiac arrhythmia, Cardiac infarction, Coronary stent / angiography, Cerebrovascular insult, Hypertension
* Pre-existing blood-borne disease: HIV, Hepatitis C, MRSA
* Pre-existing systemic or localized rheumatic illness
* Cancer
* Pre-existing psychiatric disorder
* Another pre-existing systemic disease

Ages: 45 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-30 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Compare the efficacy of the morning and afternoon HIIT in lowering blood glucose values in participants with type 2 diabetes. | 36 hours on: visit 1 (baseline / no exercise), visit 2 (Arm 1 - Morning HIIT / Arm 2 - Afternoon HIIT) and visit 3 (Arm 1 - Afternoon HIIT / Arm 2 - Morning HIIT)
  Continuous glucose monitor-based blood glucose measurements will be recorded and blood samples will be obtained before and after exercise. Additional repeated blood samples will be collected every 4-6 hours during the stay.

SECONDARY OUTCOMES:
Blood insulin levels (mIU/l) will be determined in collected blood samples and compared between exercise interventions (morning vs afternoon HIIT) as well as to no-exercise baseline measurements (morning / afternoon HIIT vs baseline). | Every 4-6 hours during 36 hours on visit 1 (baseline / no exercise), visit 2 (Arm 1 - Morning HIIT / Arm 2 - Afternoon HIIT) and visit 3 (Arm 1 - Afternoon HIIT / Arm 2 - Morning HIIT)
Respiratory exchange ratio (RER) | During exercise on visit 2 (Arm 1 - Morning HIIT (08:30) / Arm 2 - Afternoon HIIT (19:30)) and visit 3 (Arm 1 - Afternoon HIIT (19:30) / Arm 2 - Morning HIIT (08:30))
  Respiratory exchange ratio (RER) will be determined for the duration of the exercise bout utilizing a face-mask gas collector coupled to indirect calorimeter. RER comparisons will be made between the two exercise interventions (morning vs afternoon HIIT).

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided